CLINICAL TRIAL: NCT01408446
Title: A Randomized, Double-Blind, Placebo Control Trial Comparing Effects and Safety of DANSHU Capsule(Menthol) and Placebo on Blood Pressure and Metabolic Parameters in Prehypertensive and Mild Hypertensive Patients
Brief Title: Effects and Safety of Menthol on Blood Pressure and Metabolic Parameters in Prehypertensive and Mild Hypertensive Patients
Acronym: ESMAB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Chief Scientist of the National Key Basic Research and Development Program (973 Program), Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GZS01167261
Record Dates: First submitted 2011-07-25; First posted 2011-08-03 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Prehypertension
Keywords: Hypertension; Menthol; Metabolism
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Menthol (Active Comparator): Interventions Drug: Menthol Arms: Group 1
  Interventions: Drug: Menthol
- Placebo (Placebo Comparator): Interventions Drug: Placebo Arms: Group 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menthol — Capsule 48mg three times a day after meals 8 weeks
  Arms: Menthol
Drug: Placebo — Capsule 48mg three times a day after meals 8 weeks
  Arms: Placebo

SUMMARY:
Prehypertension and mild hypertension are associated with an increased risk of atherosclerosis and coronary artery disease, and often complicated with the metabolic disorder of glucose and lipid. The comprehensive prevention of hypertension is still an important and complex clinical issue. Peppermint is a popular flavoring agent, and peppermint tea help relax tension and could lower blood pressure. The effect of oral peppermint on blood pressure is not consistent, however, our previous animal study has shown that oral administration of menthol, the main component of peppermint, could reduce 24-hour mean arterial systolic and diastolic blood pressure in spontaneous hypertensive rats. Furthermore, menthol increases uncoupling protein(UCP)1 dependent thermogenesis and energy expenditure through transient receptor potential melastatin(TRPM)8 activation, and helps prevent obesity and metabolic disorders. In a prospective, double-blind, randomized, and parallel-group study, we will evaluate the effects of DANSHU capsule(menthol) on blood pressure and metabolic parameters in prehypertensive and mild hypertensive patients. This study will help develop future comprehensive prevention and treatment strategies for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure: 120mmHg≤SBP<160mmHg, and/or 80mmHg≤DBP<100mmHg

Exclusion Criteria:

* Diabetes
* Hypertension: SBP≥160mmHg, or DBP≥100mmHg
* known allergy to trial drugs
* Myocardial infarction or cerebrovascular accident in the year preceding the trial
* Clinical Congestive Heart Failure
* Secondary hypertension
* Pregnancy or lactating women
* Malignant tumor
* Gastroesophageal reflux or gastroduodenal ulcer
* History of hepatitis or cirrhosis
* History of kidney disease
* Body weight﹤35Kg

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-08-30 (Actual)

PRIMARY OUTCOMES:
The decrease in diastolic blood pressure after an 8-week oral menthol administration | 8 weeks
  Evaluate the effects of DANSHU capsule(menthol) on blood pressure and metabolic parameters in prehypertensive and mild hypertensive patients after an 8-week oral administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Sun J, Yang T, Wang P, Ma S, Zhu Z, Pu Y, Li L, Zhao Y, Xiong S, Liu D, Zhu Z. Activation of cold-sensing transient receptor potential melastatin subtype 8 antagonizes vasoconstriction and hypertension through attenuating RhoA/Rho kinase pathway. Hypertension. 2014 Jun;63(6):1354-63. doi: 10.1161/HYPERTENSIONAHA.113.02573. Epub 2014 Mar 17. PMID 24637663
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24637663